CLINICAL TRIAL: NCT03757429
Title: Inflammatory Mediators Associated With Infection by Respiratory Syncytial Virus
Acronym: IMAR
Status: Completed | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Swedish University of Agricultural Sciences (Other)
Responsible Party: Principal Investigator, Robert Frithiof, Principal Investigator, Uppsala University
Other Study IDs: 2017-515IMAR
Record Dates: First submitted 2018-11-22; First posted 2018-11-29 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Respiratory Tract Infections; Respiratory Syncytial Virus Infections
MeSH Terms: conditions — Respiratory Tract Infections; Respiratory Syncytial Virus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RS-virus infection with mechanical ventilation: Patients admitted to the pediatric ICU with verified or suspected RS-virus infection that are mechanically ventilated.
  Interventions: Other: RS-virus infection
- Non-RS-virus infection with mechanical ventilation: Patients admitted to the pediatric ICU due to a cause other than a verified or suspected respiratory tract infection.
  Interventions: Other: RS-virus infection

INTERVENTIONS:
Other: RS-virus infection — The intervention consists of lower respiratory tract infection due to RS-virus

SUMMARY:
Infection with human respiratory syncytial (RS) virus is the most common cause of hospital stay due to pediatric lower respiratory tract infection. An exaggerated immune response contributes to the pathogenesis and small children may have over reactive airways for a long time after an infection.

New research has shown that polymorphonuclear leukocytes (PMNs) are stimulated by the virus. Besides fighting the infection they also cause collateral damage to the host. Among other mechanisms PMNs stimulates mucus formation that affects breathing. They also secrete enzymes, toxic proteins and free radicals that may cause harm to lung tissue and airways.

The current project strives towards identifying and quantifying inflammatory mediators in sputum, urine and blood of children with severe RS-virus infection. The ultimate aim of the project is to, in detail, describe proteins contributing to the pathogenesis of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Admission to pediatric intensive care unit
* Clinical need for invasive ventilation
* Clinical need for intravascular catheterization
* Clinical need for urine bladder catheterization
* Patients with verified or suspected RS-virus-infection or no respiratory tract infection (control group)

Exclusion Criteria:

• Chronic inflammatory lung disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Children admitted to pediatric ICU
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Levels of inflammatory mediators in sputum | Up to three weeks
  Simultaneous detection and quantification of hundreds of potential mediators using mass-spectrometry
Levels of inflammatory mediators in blood | Up to three weeks
  Simultaneous detection and quantification of hundreds of potential mediators using mass-spectrometry
Levels of inflammatory mediators in urine | Up to three weeks
  Simultaneous detection and quantification of hundreds of potential mediators using mass-spectrometry

SECONDARY OUTCOMES:
Disease severity as measured by sequential organ failure assessment score (SOFA-score) | Up to 30-days
Lung function as measured in respirator | Up to 30-days
Lung function as measured by spirometry | Within 1 year
Lung function as measured by spirometry | Within 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Akademiska sjukhuset, Centraloperation, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No